CLINICAL TRIAL: NCT00472771
Title: A Phase II, Open-label Study of INNO-206 in Patients With Recurrent Extensive Small Cell Lung Cancer After First-line Platinum-based Therapy
Brief Title: INNO-206 in Patients With Small Cell Lung Cancer (SCLC)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to clinical trial material production delays
Sponsor: CytRx (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INNO-206-P2
Record Dates: First submitted 2007-05-11; First posted 2007-05-14 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Small Cell Lung Cancer
Keywords: Recurrent extensive small cell lung cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — DOXO-EMCH

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: INNO-206

SUMMARY:
The purpose of this study is to determine whether INNO-206 is effective in the treatment of small cell lung cancer.

DETAILED DESCRIPTION:
This is a phase II, open-label, prospective, multicenter, single-arm study of INNO 206 in adult patients with recurrent extensive small cell lung cancer sensitive to first-line platinum-based therapy. The primary objective of the study is to determine the objective overall response rate. Secondary objectives include evaluating the treatment-related toxicities in this patient population and determining the pharmacokinetic (PK) profile of INNO-206 in a minimum of 12 patients.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥18 years old.
* Have a histologically or cytologically confirmed diagnosis of recurrent extensive small cell lung cancer (SCLC) at the time of enrollment into the study.
* Have responded to first-line platinum-based chemotherapy, but progressed or relapsed ≥60 days after completion of first-line therapy.
* Have measurable disease defined by RECIST.
* Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤2.
* Have an estimated life expectancy of ≥4 weeks.
* Be male or non-pregnant, non-lactating female patients. Patients who are fertile must agree to use an effective barrier method of birth control to avoid pregnancy while on therapy and for 90 days following the discontinuation of the study medication.
* Have a negative serum or urine pregnancy test within 7 days prior to the first dose of study medication (if patient is a female of childbearing potential).
* Have adequate organ function.

Exclusion Criteria:

* Are pregnant or lactating.
* Have received prior anthracycline therapy.
* Have participated in any investigational drug study within 30 days prior to study entry.
* Have received radiotherapy within 2 weeks of treatment in this study.
* Have not recovered from acute toxicity of all previous therapy prior to enrollment.
* Have a history of a malignancy other than SCLC. Exceptions to this include: curatively treated nonmelanomatous carcinoma of the skin or in situ carcinoma of the cervix, or prior low-grade, localized prostate cancer (Gleason score ≤6); or a history of another malignancy that was curatively treated and no evidence of recurrence for a minimum of 5 years.
* Have symptomatic central nervous system (CNS) metastases.
* Have any concurrent severe or uncontrolled medical disease (such as active systemic infection, hypertension, congestive heart failure ≥NYHA Grade II, myocardial infarction within 6 months before study start, severe rhythm disturbances, etc.) that, in the opinion of the Investigator, would compromise the safety of the patient or compromise the ability of the patient to complete the study.
* Have a psychiatric disorder(s) that would interfere with consent, study participation, or follow-up.
* Have received radiotherapy with >25% involvement of the bone marrow within 6 weeks prior to study start.
* Have a known hypersensitivity to doxorubicin, 5% D-(+)-sucrose, 10 mM sodium phosphate, and/or 0.3% N-acetyltryptophane.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-05; Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
To determine the objective overall response rate (OR; complete [CR] and partial [PR] responses).

SECONDARY OUTCOMES:
To determine the rates of stable disease and progressive disease.
To determine time to progression.
To determine progression-free survival.
To determine overall survival.
To evaluate the treatment-related toxicities in this patient population.
To determine the pharmacokinetic profile of INNO-206 in a minimum of 12 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Maitland, MD, Principal Investigator — University of Chicago
Locations (7):
- United States (7):
  - University of Chicago, Chicago, Illinois
  - Billings Clinic, Billings, Montana
  - New York Oncology Hematology, P.C., Albany, New York
  - Dayton Oncology and Hematology, Kettering, Ohio
  - Signal Point Hematology/Oncology, Inc., Middletown, Ohio
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Mary Crowley Medical Research Center, Dallas, Texas